CLINICAL TRIAL: NCT01581138
Title: A Multicenter, Randomized, Open-label, Phase 2b Study to Evaluate the Efficacy and Safety of Two Regimens of All-oral Triple Therapy (VX-222 in Combination With Telaprevir [Incivek™] and Ribavirin [Copegus®]) in Treatment-Naïve Subjects With Genotype 1a Chronic Hepatitis C
Brief Title: VX-222 + Telaprevir + Ribavirin for 12 or 16 Weeks in Treatment-Naive Subjects With Genotype 1a Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VX11-222-108
Record Dates: First submitted 2012-04-17; First posted 2012-04-20 (Estimated); Last update posted 2014-07-04 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Hepatitis C Virus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — lomibuvir; telaprevir; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 12 week treatment (Experimental)
  Interventions: Drug: VX-222; Drug: telaprevir; Drug: ribavirin
- 16 week treatment (Experimental)
  Interventions: Drug: VX-222; Drug: telaprevir; Drug: ribavirin

INTERVENTIONS:
Drug: VX-222 — 400 mg tablets twice daily for oral administration
Drug: telaprevir — 1125 mg tablets twice daily for oral administration
  Other Names: VX-950, INCIVEK, INCIVO, TELAVIC
Drug: ribavirin — 1000 mg per day for subjects weighing <75 kg and 1200 mg per day for subjects weighing ≥75 kg, dosed twice daily
  Other Names: Copegus

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of two all oral regimens in subjects who have chronic hepatitis C and have not received treatment yet.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have genotype 1 chronic hepatitis C (CHC) and laboratory evidence of HCV infection for at least 6 months before the Screening Visit
* Subjects will be treatment naïve
* Subjects must have documentation of the presence or absence of cirrhosis

Exclusion Criteria:

* History or other clinical evidence of significant or unstable cardiac disease
* Evidence of hepatic decompensation
* Diagnosed or suspected hepatocellular carcinoma
* Any other cause of significant liver disease in addition to hepatitis C, which may include but is not limited to malignancy with hepatic involvement, hepatitis B, drug-or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, nonalcoholic steatohepatitis, or primary biliary cirrhosis
* History of organ transplant, with the exception of corneal transplants and skin grafts

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-07; Primary Completion 2013-06 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects who have a sustained viral response (SVR) at 12 weeks after the last planned dose of treatment | 12 weeks after the last planned dose of treatment

SECONDARY OUTCOMES:
The safety and tolerability as assessed by adverse events (AEs), vital signs, 12-lead electrocardiograms (ECGs), and laboratory assessments (serum chemistry, hematology, and urinalysis) | up to 20 weeks
The proportion of subjects who have an SVR 24 weeks after the last planned dose of the study drug | 24 weeks after the last planned dose of the study drug
The proportion of subjects who have an SVR 4 weeks after the last planned dose of the study drug | 4 weeks after the last planned dose of the study drug
The proportion of subjects who relapse (i.e., who had <lower limit of quantitation LLOQ hepatitis C virus (HCV) RNA at the end of planned study drug treatment (planned EOT) followed by ≥LLOQ HCV RNA after planned EOT) | 48 weeks either after the last planned dose of study drug or after time of failure
The proportion of subjects who achieve undetectable HCV RNA (below the lower limit of detection (< (LLOQ) undetectable) at Weeks 2, 4, 8, 12, and 16 after the first dose of study drug, and <LLOQ at the end of planned study drug treatment (planned EOT) | up to 16 weeks
Time to achieve <LLOQ undetectable HCV RNA | up to 16 weeks
The proportion of subjects who have on-treatment virologic failure defined as subjects who either have viral breakthrough or who complete the assigned treatment and have ≥LLOQ HCV RNA at the end of study drug treatment (EOT) | up to 16 weeks
The association of the interleukin-28B (IL-28B) genotype (CC versus CT versus TT) with SVR12 | 12 weeks after the last planned dose of treatment
The amino acid sequence of the nonstructural (NS)3/4A and NS5B proteins in subjects who have treatment failure | 48 weeks either after the last planned dose of study drug or after time of failure

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Vertex Pharmaceuticals Incorporated
Locations (18):
- United States (18):
  - Birmingham, Alabama
  - Anaheim, California
  - Riverside, California
  - San Diego, California
  - Englewood, Colorado
  - Orlando, Florida
  - Marietta, Georgia
  - Baltimore, Maryland
  - New York, New York
  - Asheville, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Pittsburgh, Pennsylvania
  - Germantown, Tennessee
  - Nashville, Tennessee
  - Austin, Texas
  - San Antonio, Texas
  - Norfolk, Virginia